CLINICAL TRIAL: NCT03836833
Title: Pharmacokinetic, Safety and Acceptability Study of the Abacavir/Lamivudine/Lopinavir/Ritonavir/-30/15/ 40/10mg vs. Lopinavir/Ritonavir 40/10mg Pellets Plus Dual Abacavir/Lamivudine-60/30mg Tablets in HIV Infected Children
Brief Title: Lopinavir/r/ Lamivudine/ Abacavir as an Easy to Use Paediatric Formulation
Acronym: LOLIPOP
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Drugs for Neglected Diseases (Other)
Collaborators: UNITAID (Other); AMS-PHPT Research Platform (Program for HIV Prevention and Treatment) (Unknown); Joint Clinical Research Centre- Kampala (Unknown); Baylor College of Medicine Childrens Foundation, Uganda (Unknown); Epcentre Centre Mbarara Research Centre (Unknown); Institute of Tropical Medicine, Belgium (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: DNDi-4in1-01-PHIV
Record Dates: First submitted 2018-12-13; First posted 2019-02-11 (Actual); Last update posted 2019-06-07 (Actual); Status verified 2019-05

CONDITIONS: HIV

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- 4in1 granules (Experimental): Abacavir/Lamivudine/ Lopinavir/Ritonavir (30/15/ 40/10mg ;4-in-1) Fixed-Dose Combination in granules formulation administered twice daily for at least 3 weeks, Followed by Lopinavir/Ritonavir (40/10mg pellets) plus dual Abacavir/Lamivudine (60/30mg dispersible tablets) administered twice daily for at least 3 weeks.
  Interventions: Drug: ABC/3TC/LPV/r granules (30/15/40/10 mgs); Drug: LPV/r Pellets (40/10mgs) plus ABC/3TC (60/30mgs)
- LPV/r Pellets Plus ABC/3TC (Experimental): Lopinavir/Ritonavir (40/10mg pellets) plus dual Abacavir/Lamivudine (60/30mg dispersible tablets) administered twice daily for at least 3 weeks.
  Followed by Abacavir/Lamivudine/ Lopinavir/Ritonavir (30/15/ 40/10mg ;4-in-1) Fixed-Dose Combination in granules formulation administered twice daily for at least 3 weeks
  Interventions: Drug: ABC/3TC/LPV/r granules (30/15/40/10 mgs); Drug: LPV/r Pellets (40/10mgs) plus ABC/3TC (60/30mgs)

INTERVENTIONS:
Drug: ABC/3TC/LPV/r granules (30/15/40/10 mgs) — This is a fixed dose combination. Each capsule contains Lopinavir (40mg), Ritonavir (10mg), Abacavir (30mg) and Lamivudine (15mg) in granules formulation.
  Dosage according to patient's weight:
  Between 3 and 5.9kg: 2 capsules twice a day Between 6 and 9.9kg: 3 capsules twice a day Between 10 and 13.9kg: 4 capsules twice a day Between 14 and 19.9kg: 5 capsules twice a day Between 20 and 24.9kg: 6 capsules twice a day
  Other Names: 4in1 Granules
Drug: LPV/r Pellets (40/10mgs) plus ABC/3TC (60/30mgs) — Lopinavir/Ritonavir (40/10mg pellets) plus dual Abacavir/Lamivudine (60/30mg dispersible tablets)
  Dosage according to patient's weight:
  LPV/r Pellets:
  Between 3 and 5.9kg: 2 capsules twice a day Between 6 and 9.9kg: 3 capsules twice a day Between 10 and 13.9kg: 4 capsules twice a day Between 14 and 19.9kg: 5 capsules twice a day Between 20 and 24.9kg: 6 capsules twice a day
  ABC/3TC:
  Between 3 and 5.9kg: 1 tablet twice a day Between 6 and 9.9kg: 1.5 tablets twice a day Between 10 and 13.9kg: 2 tablets twice a day Between 14 and 19.9kg: 2.5 tablets twice a day Between 20 and 24.9kg: 3 tablets twice a day
  Other Names: L PV/r Pellets Plus ABC/3TC tablets

SUMMARY:
A phase I/II, open label, randomized crossover pharmacokinetic, safety and acceptability study of the Abacavir/Lamivudine/ Lopinavir/Ritonavir (30/15/ 40/10mg ;4-in-1) Fixed-Dose Combination vs. Lopinavir/Ritonavir (40/10mg pellets) plus dual Abacavir/Lamivudine (60/30mg tablets) in HIV infected Children.

The study is intended to support the adoption of the 4-in-1 by healthcare providers and will provide data that may support its registration in certain countries. The study will be carried out in HIV-infected children in Uganda weighing 3 to 25 kg (inclusive) and unable to swallow tablets and will provide supportive clinical data on the pharmacokinetics, safety, tolerability and acceptability of the 4-in-1.

DETAILED DESCRIPTION:
The primary objective is to estimate the population average exposure to LPV, ABC and 3TC provided by the 4-in-1 formulation in HIV-infected children dosed per WHO weight bands.

The secondary objectives:

* To determine the proportion of children overall, and within each weight band, with a lopinavir C12 <1.0 mg/L while receiving the 4-in-1 formulation
* To evaluate and compare the safety and tolerability of the 4-in-1 formulation versus a reference treatment regimen.
* To compare the bioavailability of LPV, ABC and 3TC in the 4-in-1 formulation versus a reference treatment regimen.
* To assess post exposure CD4 and viral load
* To assess the factors that contribute to acceptability of the new 4-in-1 formulation.

ELIGIBILITY:
Inclusion Criteria:

* Children > 4 weeks old and weighing ≥3 and <25 kg at the time of enrolment
* Past or current documentation of a confirmed diagnosis of HIV infection defined as two positive assays from two different samples. The two results may be in any combination of the following:
* At any age: HIV-1 DNA PCR positive
* Documented past HIV-1 RNA viral load > 1,000 copies/mL plasma
* At any age >18 months of age: HIV-1 antibody reactive on two different rapid tests based on national testing algorithm
* ARV treatment eligible children with LPV-based treatment indication* as defined by country-specific guidelines or the WHO paediatric treatment guidelines and confirmed by the investigator
* HIV RNA viral load <1000 copies/mL (suppressed) at the screening visit*
* Inability to swallow LPV/r tablets
* Parent or guardian able and willing to provide written informed consent.
* For lowest weight band (≥3 and ≤ 5.9kgs) ONLY: under treatment for at least 3 weeks but not more than 12 weeks.

  * Does not apply to the youngest children (≥3 and ≤ 5.9kgs)

Exclusion Criteria:

* Planned or concurrent use of NNRTIs, integrase inhibitors, entry inhibitors, or Protease Inhibitors (PIs) other than LPV/r.
* Treatment failure with proven resistances to PIs.
* Contraindication to use of PIs
* Clinical condition requiring the use of a prohibited medication (see section 7.6) in association with LPV/r, ABC/3TC (Refer to section 7.2- 7.3 of the IB)
* Pulmonary Tuberculosis and any clinically significant disease or finding during screening that, in the investigator's opinion, would compromise participation in this study.
* Treatment with experimental drugs (except for LPV/r Pellets) for any indication within 30 days prior to study entry
* Anticipated transfer of care to a non-participating health facility during the study period

Min Age: 4 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2019-06-04 (Actual); Primary Completion 2019-11 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
0 -12 hours Area under the curve plasma concentration versus time for LPV, ABC and 3TC in the 4-in- formulation | 0-12 hours
  0 -12 hours Area under the curve plasma concentration versus time for LPV, ABC and 3TC in the 4-in- formulation

SECONDARY OUTCOMES:
Plasma concentration at 12 hours for LPV in the 4in1 formulation | 12 hours
  Plasma concentration at 12 hours for LPV in the 4in1 formulation
Peak plasma concentration (Cmax) of LPV, ABC and 3TC with the 4-in-1 formulation. | 3-5 weeks
  Plasma concentration maximum of LPV, ABC and 3TC with the 4-in-1 formulation.
Concentration time maximum for LPV, ABC and 3TC with the 4-in-1 formulation. | 3-5 weeks
  Concentration time maximum for LPV, ABC and 3TC with the 4-in-1 formulation.
Clearance function for LPV, ABC and 3TC with the 4-in-1 formulation. | 3-5 weeks
  Clearance function for LPV, ABC and 3TC with the 4-in-1 formulation.
Geometric mean ratio (GMR) of steady state LPV, ABC and 3TC versus time (0-12) in the 4-in-1 formulation versus the reference treatment regimen | 0 - 12 hours
  Geometric mean ratio (GMR) of steady state LPV, ABC and 3TC versus time (0-12) in the 4-in-1 formulation versus the reference treatment regimen.
Area under curve plasma concentration versus time (0-12) in the 4-in-1 formulation versus the reference treatment regimen. | 0 - 12 hours
  Area under curve plasma concentration versus time (0-12) in the 4-in-1 formulation versus the reference treatment regimen.
Geometric mean ratio (GMR) of steady state LPV, ABC and 3TC in the 4-in-1 formulation versus the reference treatment regimen. | 0 - 12 hours
  Geometric mean ratio (GMR) of steady state LPV, ABC and 3TC in the 4-in-1 formulation versus the reference treatment regimen.
Peak plasma concentration in the 4-in-1 formulation versus the reference treatment regimen. | 3-5 weeks
  Peak plasma concentration in the 4-in-1 formulation versus the reference treatment regimen.
Safety: A description of the proportion of children experiencing an Adverse event or Serious Adverse event binomial distribution compared between the two formulations. | 6-8 weeks
  Safety: A description of the proportion of children experiencing an Adverse event or Serious Adverse event binomial distribution compared between the two formulations.
Safety: Summary of the number and percent of subjects with documented Grade 3 or higher adverse events; each summary will be conducted overall and by formulation | 6-8 weeks
  Safety: Summary of the number and percent of subjects with documented Grade 3 or higher adverse events; each summary will be conducted overall and by formulation
Proportion of children with viral load <1000 copies/ml | 6-8 weeks
  Comparison of proportion of children with viral load less than 1000 copies/ml at baseline and at end of the study.
Changes in CD4 counts compared to baseline | 6-8 week
  Changes in CD4 counts compared to baseline
Changes in CD4 percentage compared to baseline | 6-8 weeks
  Changes in CD4 percentage compared to baseline
Acceptability: Description of factors that affect acceptability of the 4 in1 formulation | 6-8 weeks
  Description of factors that affect acceptability of the 4in1 formulation as reported by the caregivers

CONTACTS AND LOCATIONS:
Overall Officials: Isabelle Andrieux-Meyer, MD, Study Director — Drugs for Neglected Diseases initiative
Locations (3):
- Uganda (3):
  - Baylor College of Medicine Children's Foundation Uganda, Kampala
  - Joint Clinical research Centre, Kampala
  - Epicentre Mbarara Research Centre, Mbarara

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Rotsaert A, Ogara C, Mwanga-Amumpaire J, Kekitiinwa AR, Musiime V, Najjingo E, Kisitu GP, Nazzinda R, Nambi E, Lee J, Diallo M, Kyomuhendo F, Waweru M, Andrieux-Meyer I, Nostlinger C. Acceptability of a new 4-in-1 Abacavir/Lamivudine/Lopinavir/Ritonavir paediatric fixed-dose combination: the caregiver-child dyads' perspective. Ther Adv Infect Dis. 2023 Mar 21;10:20499361231159993. doi: 10.1177/20499361231159993. eCollection 2023 Jan-Dec. PMID 36968554